CLINICAL TRIAL: NCT05885893
Title: The Effect of Smartphone Addiction Level on Neck Pain, Functional Status and Muscle Activation
Brief Title: Smartphone Addiction Level and Neck Muscle
Status: Completed | Type: Observational
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Menekse Safak, Principal Investigator, Suleyman Demirel University
Other Study IDs: MS2022/033
Record Dates: First submitted 2023-04-18; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Smartphone Addiction; Neck Muscle Issue
Keywords: Smartphone Addiction; Neck Muscles; Pain; Muscle Activation; Functional Status
MeSH Terms: conditions — Internet Addiction Disorder; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background/aim:The study was conducted to determine the smartphone addiction level of youths and to investigate the effect of addiction level on neck pain, functional level, pressure pain threshold (PPT) level, and muscle activation of neck muscles (upper trapezius (UT), cervical erector spina (CES), sternocleidomastoideus (SCM)).

Methods:Superficial electromyography, PPT, Visual Analog Scale (VAS), Neck Disability Index (NDI) and Smartphone Addiction Scale (SAS) were used as assessment tools.

DETAILED DESCRIPTION:
Smartphones, which are used quite frequently among adolescents, are becoming more and more indispensable in daily life and offer a wide variety of mobile applications for information, communication, education, and entertainment. The use of smartphones includes many user profiles such as teenagers, adults, children, working or not working. However, when looking at the smartphone user profile, it is seen that the largest proportion belongs to the young population.

With the increasing frequency of use and addiction, many physiological, psychological, and social problems are encountered today. These problems can be classified into two categories that are psychological disorders (sleep disorders, aggressive or depressive symptoms, high anxiety level, low life satisfaction, dropping out of school, and antisocial personality disorder) and physiological disorders (dry eyes, carpal tunnel syndrome, neck or back pain, postural disorders, musculoskeletal disorders, and migraine headaches). Regarding its adverse effects on physical health, especially the increase in neck pain and the decrease in daily life activities and functionality are emphasized. The effects of smartphone use on the functional level are associated with the cervical posture and the sensitivity, spasm and proprioceptive disorders in the neck circumference structures created by this posture. Smartphone addiction and computer addiction, which has similar effects, are associated with neck problems and disability in healthy young people. It has been reported that smartphone addiction in students negatively affects physical health by reducing the amount of physical activity such as walking. In the literature, an increase in muscle fatigue and increased sensitivity in cervical erector spina (CES) and upper trapezius (UT) muscles have been reported due to prolonged smartphone use. Although there are data on the negative effects of smartphone use on many physiological parameters such as pain and functional level in the literature, there is a need for studies evaluating the effect of smartphone addiction, which has emerged as an important concept in recent years.

Posture during phone use stands out as the primary cause of musculoskeletal disorders associated with smartphone use. During the use of the smartphone, the person maintains the posture in which the head is in flexion and the shoulder is in protraction for a long time to look at the device. It is known that the loads on the neck increase with the flexion of the head. This situation has effects not only on the neck musculoskeletal system but also on the shoulder and spine as it creates muscle imbalance. In current studies, it has been emphasized that posture disorder during smartphone use changes the activity of the UT muscle, CES muscle, neck extensor muscles, and hand muscles.

There are various studies in the literature on muscle activation changes, musculoskeletal system changes, and changes in daily living activities with the use of smartphones. However, it is thought that there is a need for a study that correlates smartphone addiction with musculoskeletal problems such as pain and sensitivity, muscle activation changes in the neck muscles, and changes in functional status. It is thought that the determination of physiological effects such as neck pain and muscle activations that they cause even when they do not use phones, even when they do not use telephone, are thought to be effective in terms of drawing attention to the importance of preventing them. In light of this information, our study aimed to examine the effect of smartphone addiction levels on neck pain, functional status, and muscle activation.

ELIGIBILITY:
Inclusion Criteria:

* to be studying at Süleyman Demirel University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation,
* volunteering to participate in the study,
* for the past 6 months, using a smartphone for at least 2 hours a day.

Exclusion Criteria:

* a history of surgical intervention or traumatic injury in the spine and upper extremity,
* chronic disease affecting the musculoskeletal system such as rheumatoid arthritis, osteoarthritis and other connective soft tissue diseases,
* sensory impairment in the spine or upper extremities to have a neurological and orthopedic disorder,
* activities such as long-term reading, which will affect the flexion posture of the head, have been performed in the last 1 month,
* having done exercises involving neck muscles in the last 1 month.

Ages: 15 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: A total of 112 male university students studying at Süleyman Demirel University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation were included in study.
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2017-12-10 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Neck Pain Intensity Assessment | 1 month
  The Visual Analogue Scale (VAS) was used to evaluate the neck pain intensity. VAS is a continuous scale, it is a horizontal line of 100 mm in length, anchored by 2 adjectives: zero representing no pain in the left anchor and 10 representing worst imaginable pain at the right anchor. The participant was asked to mark the point corresponding to the intensity of pain felt on this line. The numerical value found indicates the pain severity of the participants.
Smartphone Addiction Level Assessment | 1 month
  The smartphone addiction level was assessed by Smartphone Addiction Scale (SAS). The assessment of validity and reliability of its Turkish version in a younger population was performed. SAS is a suitable tool for assessing smartphone addiction in younger population. The scale consists of 7 factors that evaluate daily life disturbance and tolerance (1. factor), withdrawal symptoms (2. factor), positive expectation (3. factor), cyber-oriented relationships (4. factor), excessive use (5. factor), social network addiction (6. factor) and physical symptoms (7. factor). The scores on the scale can range from 33 to 198. High score indicating a more serious smartphone addiction level.
Functional Level Assessment | 1 month
  Functional level was assessed by the Neck Disability Index (NDI). The assessment of validity and reliability of its Turkish version was performed. Survey questions; Daily life activities such as lifting, working, driving, resting consist of 4 titles, optional activities in daily life such as personal care consist of 2 titles, and subjective symptoms such as pain sensitivity, headache, concentration, sleep consist of 4 titles. The highest score is 50 and the lowest score is 0. Classification by total score; 0-4 points no disability, 5-14 points mild disability, 15-24 points moderate disability, 25-34 points severe disability, 34 points and above completely disability. The participants were asked to answer the questions based on the neck pain they felt during the past 1 week.
Pain Sensitivity Level Assessment | 1 month
  Pressure pain threshold (PPT) is used to assess sensitivity to pain and pressure perception. Using a Wagner Instruments, Force Dial (TM FDK/FDN, Greenwich, CT, USA) device, a constant force of 1 kg / cm2 was applied to the CES, UT and SCM muscles bilaterally. The pressure pain threshold measurement at each site was repeated three times and the average of the three repetitions was used for further analysis. Participants rested for 5 minutes between each measurement.
Muscle Activation Level Assessment | 1 month
  The activation of neck muscles consisting of SCM, UT and CES muscles were measured by surface electromyography (sEMG). Measurements were made in the resting position bilaterally. For the resting position, the patient was evaluated in a chair without back support, in a sitting position with arms supported in front, and a posture without pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Menekşe ŞAFAK, Merkez, Isparta, Turkey (Türkiye)